CLINICAL TRIAL: NCT04972890
Title: The Outcomes of Intracavernosal Umbilical Cord Mesenchymal Stem Cells Implantation in Patients With Diabetic Erectile Dysfunction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Gampo Alam Irdam, Lecturer, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-04-0516
Record Dates: First submitted 2021-07-06; First posted 2021-07-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Urologic Diseases; Erectile Dysfunction With Diabetes Mellitus
MeSH Terms: conditions — Urologic Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): with 2cc saline/NaCl 0,9% solution once at baseline
  Interventions: Other: placebo
- Stem Cell Group (Experimental): with umbilical cord stem cells 15x10^6 cells in 2 cc saline/NaCl 0,9% solution once at baseline
  Interventions: Biological: stem cells

INTERVENTIONS:
Biological: stem cells — Using umbilical cord stem cells 15x10^6 cells in 2 cc saline/NaCl 0,9% solution
  Arms: Stem Cell Group
Other: placebo — using 2 cc saline/NaCl 0,9% solution
  Arms: Control group

SUMMARY:
Erectile dysfunction (ED) is a complex condition affecting men worldwide. Diabetes mellitus (DM) is one of the most common causes of ED. The prevalence of ED in DM varies around 35-85%. Recently, stem cell therapy has started to become the focus of experimental and clinical studies for the treatment of ED. Stem cells have been shown to be able to regenerate functionally damaged tissue, depending on the stimuli or signals received. Stem cells studies in experimental animals have been carried out using biomarker parameters, including VEGF, Bcl-2, E-selectin, cGMP, eNOS and have been shown to be successful in increasing cell survival and angiogenesis, stimulating antiapoptotic, proneurogenic, proinflammatory, and antifibrotic effects and improvements to these biomarker parameters. This study aims to determine the efficacy, mechanism of action, and safety of umbilical cord mesenchymal stem cells as a therapy for ED due to type 2 diabetes in human.

DETAILED DESCRIPTION:
Prior to conducting clinical trials, researchers asked for written informed consent. If the subject agrees, the study will direct the subject and control to collect basic data in the form of vital signs, blood pressure, filling out the IIEF-5 questionnaire, complete blood count (CBC), lipid profile, fasting blood glucose, HbA1c, and total testosterone, biomarker examination (E-Selectin), VEGF, Bcl-2, miRNA 16, miRNA 126), and penile Doppler ultrasound. The diagnosis of erectile dysfunction was made on the basis of an IIEF-5 score <22.

Penile Doppler ultrasound was performed by a senior radiologist with interpretation of the ultrasound images performed and reported in a blinded fashion (the reader/interpreter does not know the patient's complaints). Penile Doppler ultrasound examination was performed under flaccid conditions and post-sexual stimulation conditions. Prior to the examination, the patient was given sildenafil 100 mg orally, then the flaccid phase was examined. Patients were asked to perform sexual stimulation of themselves and measurements were taken afterwards.

Parallel with the patient recruitment, stem cells processing was carried out based on the production method using xeno-free material.

At the baseline, patient receive intracavernous injection procedure, as a following steps:

* The base of the penis is clamped with ethiloop before the injection is performed.
* Intracavernous injection was performed in each body of 7.5 x 10^6 cells/1cc.
* Clamps are removed after 30 minutes post-injection to increase stem cell residency and grafting time.

After the procedure, we monitor the symptoms for 1 hour to assess the presence or absence of complications before the subject can go home.

We also administer PDE-5 inhibitor to all research subjects, namely tadalafil at a dose of 1 x 2.5 mg for 3 months.

Follow-up was carried out on all subjects both from the experimental group and the control group by evaluating parameters consisting of IIEF-5, DPL, Lipid profile, HbA1c, GDS, total testosterone, Doppler ultrasound, e-selectin, Bcl-2, VEGF, miRNA 16, miRNA 126 at first and third month after baseline.

After all data have been collected, we will perform data analysis and make research report.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old
* willing to participate as research subject
* patient with erectile dysfunction and Diabetes Mellitus type 2 with IIEF-5 score <22
* patient has sexual partner and sexually active
* patient is currently not consuming PDE-5 inhibitor drugs

Exclusion Criteria:

* patient has psychopathology and/or mental retardation
* patient with Peyronie's disease
* patient with hypogonadism
* patient has malignancy in urological and non urological fields
* patient has history of cardiovascular disease with intermediate and high risk

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in IIEF-5 Score after stem cells injection | The questionnaire will be completed at baseline, 1st month, and 3rd month
  using IIEF-5 Questionnaire [numeric scale from 0 to 25] higher IIEF-5 Score means better erectile function
Changes in Peak Systolic Velocity (PSV) after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by penile doppler ultrasound [ numeric scale in cm/s] The normal value is 35cm/s, PSV <35cm/s means worse erectile function
Changes in End Diastolic Velocity after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by penile doppler ultrasound [ numeric scale in cm/s] The normal value is 5 cm/s, EDV >5cm/s means worse erectile function
Changes in Resistive Index after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by penile doppler ultrasound [numeric scale] The normal value is >0.9, if RI<0.75 means worse erectile function
Changes in Pulsatility Index after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by penile doppler ultrasound [numeric scale]
Changes in E-selectin expression after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by biomolecular examination using blood sample [numeric scale]
Changes in Vascular Endothelial Growth Factor (VEGF) expression after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by biomolecular examination using blood sample [numeric scale]
Changes in Bcl-2 expression after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by biomolecular examination using blood sample [numeric scale]
Changes in microRNA 16 expression after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by biomolecular examination using blood sample [numeric scale]
Changes in microRNA 126 expression after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  evaluated by biomolecular examination using blood sample [numeric scale]

SECONDARY OUTCOMES:
Changes in Hba1c after stem cells injection | The evaluation will be completed at baseline and 3rd month
  using blood sample [numeric scale in %]
Changes in Fasting Blood Glucose after stem cells injection | The evaluation will be completed at baseline and 3rd month
  using blood sample [numeric scale in mg/dL]
Changes in total cholesterol after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  using blood sample [numeric scale in mg/dL]
Changes in low-density lipoprotein (LDL) after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  using blood sample [numeric scale in mg/dL]
Changes in high-density lipoprotein (HDL) after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  using blood sample [numeric scale in mg/dL]
Changes in Triglycerides (TG) level after stem cells injection | The evaluation will be completed at baseline, 1st month, and 3rd month
  using blood sample [numeric scale in mg/dL]
Number of participants with side effects after intracavernosal injection | The evaluation will be completed at baseline after the injection
  To evaluate the number of participants with side effects including: pain, swelling, bleeding, hypesthesia, and voiding difficulty after the injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia